CLINICAL TRIAL: NCT06366308
Title: Decade-Long Insights Into Transperineal Prostate Biopsy in a West China Population: Temporal Trend, Targeted and Repeat Biopsies, and Pathological Characterization: Comparative Study - Retrospective Cohort
Brief Title: Decade-Long Insights Into Transperineal Prostate Biopsy in a West China Population
Status: Not yet recruiting | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Hao Zeng, Professor, West China Hospital
Other Study IDs: ProBiox
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Prostate Cancer; Pathology
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Transperineal Prostate Biopsy — The investigators plan to retrospectively review data from over 10000 men receiving transperineal prostate biopsy in our center.

SUMMARY:
Prostate cancer (PCa) remains one of the most prevalent malignancies affecting men globally. The disease spectrum of PCa ranges from indolent tumors, which may require minimal to no intervention, to aggressive, potentially lethal forms. The complexity of PCa underscores the critical need for precise diagnostics, as early and accurate detection is key to improving patient outcomes and tailoring appropriate treatment strategies. There have been remarkable advancements in biopsy technology. Significant strides in magnetic resonance imaging (MRI), especially with the establishment of the Prostate Imaging Reporting and Data System (PI-RADS), have substantially improved the accuracy of PCa detection. The combination of MRI with traditional biopsy methods, including MRI-targeted biopsy (MRI-TBx) and systematic biopsy (SBx), also marks a major advancement in the field.

Despite advances in PCa detection, the need for improving diagnostics and in-depth assessment of the latest PBx techniques through extensive, longitudinal studies remains critical. Besides, based on the world health organization (WHO) classification, PCa includes a range of pathological forms beyond the commonly known acinar adenocarcinoma. However, the prevalence and demographic distribution of non-adenocarcinoma types, as well as the characteristics of patients with these rarer forms, remain unclear. Leveraging PBx records spanning over 10 years and involving 10,038 cases, this study aims to shed light on temporal trends in PBx positivity, the evolving clinical profiles of PCa patients, and the differences in clinicopathological characteristics of PCa between Western and Asian populations.

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected of PCa who underwent transperineal PBx at our medical center, from 2011 to 2022

Exclusion Criteria:

* Patients with other cancers

Ages: 40 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective study analyzed data from 10,038 patients suspected of PCa who underwent transperineal PBx at our medical center, from 2011 to 2022.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Positive rate of prostate biopsy | 10 Years
  The investigators intend to analyze the variation in the positivity rate of prostate biopsies over several years.

IPD SHARING:
Plan to Share IPD: Undecided